CLINICAL TRIAL: NCT01726205
Title: Perioperative Pregabalin and Continuous Wound Infusion for Pain Control Following Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Sidiropoulou Tatiana, Lecturer in Anesthesiology, University of Athens, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRGCWI1
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Post-thoracotomy Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- pregabalin (Active Comparator): perioperative pregabalin starting the evening before surgery, and for five days postoperatively
  Interventions: Drug: Pregabalin and normal saline infusion, PRG
- pregabalin and continuous wound infusion (Active Comparator): Pregabalin as previous group and continuous infusion of ropivacaine 0.2% via a wound catheter
  Interventions: Drug: Pregabalin and ropivacaine 02% infusion
- placebo (Placebo Comparator): Placebo drug and normal saline infusion
  Interventions: Drug: Placebo drug, normal saline infusion

INTERVENTIONS:
Drug: Pregabalin and normal saline infusion, PRG
  Arms: pregabalin
Drug: Pregabalin and ropivacaine 02% infusion
  Arms: pregabalin and continuous wound infusion
Drug: Placebo drug, normal saline infusion
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the efficacy of pregabalin or pregabalin and continuous wound infusion versus placebo for analgesia following thoracotomy

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for a thoracotomy,

Exclusion Criteria:

* age >70 years
* BMI > 30
* preoperative Hb < 10 mg/dL
* preexistent chronic pain
* neurologic disease
* chronic assumption of alcohol
* treatment with analgesics, anxiolytics, sedatives, antidepressants, or calcium channel inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pain control | 5 days postoperatively

SECONDARY OUTCOMES:
morphine consumption | 3 days postoperatively

OTHER OUTCOMES:
side effects, pain at 1 and 3 months, incidence of neuropathic pain | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Sidiropoulou, Principal Investigator — Attikon Hospital; Eyaggelos Giavasopoulos, Principal Investigator — Attikon Hospital
Locations (1):
- Attikon Hospital, Athens, Greece